CLINICAL TRIAL: NCT01985022
Title: Autism Center of Excellence: Project 3 - Changing Developmental Trajectories Through Early Treatment
Brief Title: Changing Developmental Trajectories Through Early Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant enrollment was hindered by the COVID-19 pandemic and the study was ultimately terminated.
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nathan A. Call, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00064779; P50MH100029 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-15 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorders
Keywords: autism; pervasive developmental disorders; toddlers; behavioral intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-ESI (Active Comparator): Infants 12 months of age at risk of developing ASD who are randomized to receive the Group-ESI intervention for 9 months.
  Interventions: Behavioral: Group-ESI
- Individual-ESI plus Group-ESI (Experimental): Infants 12 months of age at risk of developing ASD who are randomized to receive Individual-ESI intervention in addition to the Group-ESI intervention for 9 months.
  Interventions: Behavioral: Group-ESI; Behavioral: Individual-ESI

INTERVENTIONS:
Behavioral: Group-ESI — The Group-ESI intervention consists of weekly small group meetings where families receive information about social communication, emotional regulation, play development, and behavioral challenges in toddler playgroups in a relaxed, supportive, child-friendly setting that provides the opportunity to talk with a professional and meet other parents.
Behavioral: Individual-ESI — The Individual-ESI intervention consists of twice-weekly home-based individualized coaching sessions. Parents learn how to support their child's communication, social, and play skills in everyday routines, activities, and places. Individual-ESI begins with an initial home visit, followed by a month of program planning, 6 months of intervention implementation, and 2 months of generalization. During generalization, the clinician meets with the family in a variety of community settings to teach the parent how to implement strategies in new settings.
  Arms: Individual-ESI plus Group-ESI

SUMMARY:
The major objective of this research protocol is to directly compare two parent intervention conditions of Early Social Interaction (ESI) for 9 months on developmental trajectories of infants showing early risk for Autism Spectrum Disorder (ASD). Participants will be randomized to receive an information, education and support group (Group) ESI intervention offered weekly, or a parent-implemented intervention (Individual) ESI intervention offered in twice-weekly, in combination with the Group ESI intervention.

DETAILED DESCRIPTION:
Mounting evidence exists of the effectiveness of intensive early intervention for a substantial proportion of children with autism spectrum disorders (ASD). Furthermore, age of entry into intervention may be predictive of outcome. Children with ASD in intensive interventions beginning by 3.5 years of age had significantly better outcomes than those beginning after age 5. These findings support the importance of early identification and intervention for improving outcomes. There is very limited research on children with ASD under 3 years of age primarily because the median age for diagnosis in the US is 5.5 years. With advances in earlier screening and diagnosis, there is a pressing need to develop early intervention programs that are appropriate and effective with very young children with ASD.

The Early Social Interaction (ESI) Project is an intervention program developed for toddlers at risk for ASD and their families as a model demonstration project funded by the United States Department of Education. ESI was designed to incorporate the National Research Council (NRC) recommendations within the context of a family-centered, natural-environments approach. The major components of ESI are:

1. routines-based intervention in natural environments
2. individualized curriculum
3. parent-implemented intervention

The Emory Autism Center of Excellence (ACE) will recruit parent-infant dyads at 12 months of infant's age from a pool of "High-Risk for Developing ASD" younger siblings and from a pool of low risk infants being studied at the Emory ACE. Parents are involved in the intervention itself while the study outcome measures are focused on the infants that are receiving the different interventions (demographic and outcome data are not collected on the parents of the infants). Infant participants will be randomized to receive an ESI intervention delivered in a group setting, or an individual ESI intervention combined with the group ESI. The intervention will last 9 months and infants will be followed until they reach 36 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Participants are recruited from the Emory Autism Center of Excellence Center from a pool of younger siblings who are at high or low risk of developing ASD
* For high-risk infants, a positive screen on 2 of 4 screening measures indicating the presence of diagnostic features of ASD by 12 months of age
* For low-risk infants will be a positive screen on 3 of 4 screening measures
* Families agree to twice monthly play group sessions for 9 months and 2-3 intervention sessions per week for 9 months (usually within work-day hours)

Exclusion Criteria:

* none

Ages: 9 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Call, PhD, Principal Investigator — Emory University, Marcus Autism Center, Children's Healthcare of Atlanta; Amy Wetherby, Ph.D., Study Director — Florida State University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Marcus Autism Center in Atlanta, Georgia, USA. Participant enrollment began in May 2013 and follow-up was completed by November 26, 2019.
Pre-assignment Details: Infants were enrolled with a parent as parents were a necessary part of the intervention that the infants received. Parents are not considered to be participants who received a study intervention, thus, only infants are described in the modules for Participant Flow, Baseline Characteristics, Outcome Measures, and Adverse Events.
Groups:
- Group-Early Social Interaction (ESI): Infants 12 months of age at risk of developing autism spectrum disorders (ASD) who were randomized to receive the Group-Early Social Interaction (ESI) intervention for 9 months
- Individual-ESI Plus Group-ESI: Infants 12 months of age at risk of developing ASD who were randomized to receive Individual-ESI intervention in addition to the Group-ESI intervention for 9 months.
Period: Overall Study
Arm/Group | Group-Early Social Interaction (ESI) | Individual-ESI Plus Group-ESI
Started | 16 | 17
Completed | 12 | 14
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group-ESI: Infants 12 months of age at risk of developing ASD who were randomized to receive the Group-ESI intervention for 9 months
- Total: Total of all reporting groups
Arm/Group | Group-ESI | Individual-ESI Plus Group-ESI | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 17 | 33
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 12 | 11 | 23
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Communication and Symbolic Behavior Scales (CSBS) Score
Description: Social communication skills were measured with the Communication and Symbolic Behavior Scales (CSBS) Behavior Sample. Interactions between the child and caregiver were videotaped and later converted to scores. The standardized total score has a mean of 100 and standard deviation of 15. Scores below 100 indicate below average performance with the social, speech, and symbolic composites.
Time Frame: Baseline (12 months of age, prior to treatment), 15, 21, and 24 months of age
Population: This analysis includes participants remaining in the study at the indicated time point who also completed this assessment. Due to scheduling conflicts with families, not all participants were able to complete every study assessment. If a study visit could not be scheduled within the visit window then that visit was skipped and the next assessment was scheduled.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group-ESI | Individual-ESI Plus Group-ESI
Number analyzed (Participants) | 16 | 17
score on a scale
  Baseline (12 months of age, prior to treatment) | 80.44 (3.83) | 78.71 (5.97)
  15 Months of Age: number analyzed (Participants) | 15 | 14
  15 Months of Age | 79.20 (10.88) | 80.36 (8.64)
  21 Months of Age: number analyzed (Participants) | 10 | 10
  21 Months of Age | 85.60 (12.85) | 91.20 (11.81)
  24 Months of Age: number analyzed (Participants) | 14 | 13
  24 Months of Age | 85.79 (17.48) | 89.92 (15.10)

2. Primary Outcome: Autism Diagnostic Observation Schedule (ADOS) Score
Description: Autism symptoms were measured with the Autism Diagnostic Observation Schedule, Second Edition which is the best gold standard diagnostic measure of ASD. The revised algorithms forming Social-Affect and Restricted Repetitive Behavior ratings of autism symptoms were used. A total of score of 1 to 3 indicates no signs of autism, a score of 4 or 5 suggests that the child may have autism spectrum disorder, while a score of 6 to 10 is indicative of autism.
Time Frame: 15, 24, and 36 months of age
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group-ESI | Individual-ESI Plus Group-ESI
Number analyzed (Participants) | 16 | 16
score on a scale
  15 Months of Age | 3.88 (2.03) | 3.75 (2.24)
  24 Months of Age: number analyzed (Participants) | 14 | 13
  24 Months of Age | 5.14 (2.69) | 5.23 (3.00)
  36 Months of Age: number analyzed (Participants) | 14 | 15
  36 Months of Age | 3.79 (2.12) | 4.53 (3.56)

3. Primary Outcome: Mullen Scales of Early Learning (MSEL) Score
Description: The Mullen Scales of Early Learning (MSEL) measures developmental level with standardized scores in five domains: Visual Reception, Receptive Language, Expressive Language, Fine Motor Skills, and Gross Motor Skills. Domain scores are represented in T-scores, with a mean of 50 and standard deviation of 10. A Verbal Composite score is calculated by averaging T-scores of the domains for Receptive and Expressive Language. A Nonverbal Composite score is calculated by averaging T-scores for Visual Reception and Fine Motor domains. Scores below 50 indicate below average performance.
Time Frame: Baseline (12 months of age, prior to treatment), 24, and 36 months of age
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Group-ESI | Individual-ESI Plus Group-ESI
Number analyzed (Participants) | 16 | 17
t-score
  Baseline (12 months of age, prior to treatment) - Verbal Composite Score | 37.50 (8.43) | 37.03 (6.16)
  24 Months of Age - Verbal Composite Score: number analyzed (Participants) | 14 | 13
  24 Months of Age - Verbal Composite Score | 40.86 (14.20) | 45.19 (11.02)
  36 Months of Age - Verbal Composite Score: number analyzed (Participants) | 15 | 15
  36 Months of Age - Verbal Composite Score | 44.43 (12.94) | 43.63 (11.73)
  Baseline (12 months of age, prior to treatment) - Nonverbal Composite Score | 54.13 (5.66) | 52.79 (8.78)
  24 Months of Age - Nonverbal Composite Score: number analyzed (Participants) | 14 | 13
  24 Months of Age - Nonverbal Composite Score | 52.36 (6.34) | 47.19 (10.70)
  36 Months of Age - Nonverbal Composite Score: number analyzed (Participants) | 15 | 15
  36 Months of Age - Nonverbal Composite Score | 48.93 (13.73) | 47.13 (10.17)

4. Primary Outcome: Vineland Adaptive Behavior Scales, Second Edition (Vineland II) Score
Description: The Vineland II assesses adaptive behavior by providing a standard score in four domains of Communication, Daily Living Skills, Socialization, and Motor Skills. Domain scores and the Adaptive Behavior Composite score are standardized with a mean of 100 with a standard deviation of 15. Scores less than 100 indicate below average performance.
Time Frame: Baseline (12 months of age, prior to treatment), 24, and 36 months of age
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group-ESI | Individual-ESI Plus Group-ESI
Number analyzed (Participants) | 16 | 16
score on a scale
  Baseline (12 months of age, prior to treatment) | 87.69 (8.51) | 87.19 (7.26)
  24 Months of Age: number analyzed (Participants) | 11 | 7
  24 Months of Age | 90.64 (8.91) | 92.14 (7.08)
  36 Months of Age: number analyzed (Participants) | 8 | 7
  36 Months of Age | 90.13 (10.75) | 84.57 (6.21)

5. Other Pre Specified Outcome: Expressive Language Phase
Description: The child's expressive language phase will be determined at each assessment based on the benchmarks delineated by Tager-Flusberg and colleagues and recommended for evaluating the efficacy and comparing outcomes across NIH-funded intervention studies. Based on multiple sources of information about language benchmarks, the language will be categorized as: Preverbal Communication, First Words, Word Combinations, or Sentences, to provide a clinically meaningful measure of language outcome.
Time Frame: Baseline (12 months of age, prior to treatment), 15, 21, 24, and 36 months of age
Population: Expressive language phase was to be coded based on the CSBS, however, this coding requires extensive time and effort by a trained staff member. As the study terminated early and research priorities shifted with the Coronavirus disease 2019 (COVID-19) pandemic, staffing was no longer available to review the video recordings specifically to code language phase. Data analyses for this study focused on addressing the primary aims of the study and data for this outcome were never created.
Arm/Group | Group-ESI | Individual-ESI Plus Group-ESI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment (up to 36 months of age).
Arm/Group | Group-ESI | Individual-ESI Plus Group-ESI
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT01985022/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT01985022/ICF_001.pdf